CLINICAL TRIAL: NCT04415281
Title: Photobiomodulation for the Management of Temporomandibular Disorder Pain
Acronym: PBM
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding not secured
Sponsor: University of Florida (Other)
Collaborators: National Institute of Dental and Craniofacial Research (NIDCR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: IRB202000766
Record Dates: First submitted 2020-04-15; First posted 2020-06-04 (Actual); Results first posted 2023-10-12 (Actual); Last update posted 2023-10-12 (Actual); Status verified 2023-10

CONDITIONS: Pain Related to TMD

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (2):
- Active PBM (Experimental): PBM has been used clinically in the treatment of musculoskeletal and other pain conditions for over 30 years. Despite the low quality of the existing evidence, PBM has been increasingly used in other countries for the treatment of TMD. However, in the US PBM is not widely used for the treatment of TMD pain. Due to the multifactorial nature of chronic TMD pain, we propose that a multimodal PBM protocol targeting multiple pathophysiological mechanisms will be the optimal approach for PBM implementation in patients with TMD.
  Interventions: Device: THOR® laser system
- Sham PBM (Sham Comparator): When applying PBM therapy, there are some heating elements in the treatment device, and most of the sham treatment devices available do not offer this feature, which increases the likelihood of unblinding both the patient and the interventionist. The THOR® LX2.3 PBM machine includes this new feature, such that the sham condition mimics the heating activity of the active treatment.
  Interventions: Device: sham THOR® laser system

INTERVENTIONS:
Device: THOR® laser system — We chose the THOR® laser system given because their active treatment arm uses both coherent laser and monochromatic LED light. Therefore, we will use three types of active probes in this investigation including, A) Single Laser 810 NM 200 mw; B) Laser Cluster of 810 NM equivalent to 1 WATT and; C) LED Cluster, 34 X 660nm at 10 mw and 35 850nm, 30mw 1390mw total. As detailed in Table 3. We propose to use these three PBM probes in concert for the treatment of TMD pain. Laser A (Single Diode Laser) is designed for isolated trigger points and superficial muscles. Laser B (Cluster Laser) is designed for a more diffuse treatment area,targeting analgesia, anti-inflammatory, and deep tissue repair. Laser C (LED Cluster) is purportedly designed for the presence of diffuse inflammation.
  Arms: Active PBM
Device: sham THOR® laser system — sham THOR® laser system
  Arms: Sham PBM

SUMMARY:
Photobiomodulation (PBM), is FDA-approved for temporary relief of muscle and joint pain, but there is no indication for TMD. Our goal in this study is to conduct a clinical trial of multimodal PBM for TMD pain. Also, we propose to determine if PBM-induced changes in inflammation contribute to PBM's analgesic effects. This study will be a double-blind, sham-controlled, randomized trial testing the efficacy of PBM for pain related to TMD.

ELIGIBILITY:
Inclusion Criteria:

* Provides a signed and dated informed consent form
* Is at least 18 years of age (male or female and any race or ethnicity)
* Meets diagnostic criteria for TMD, ( Masticatory Muscle Disorders, 1A: Myalgia)
* Has experienced facial pain for at least 3 months
* At Screening and Baseline Visit (Visit 0), reports an average pain intensity rating over the past week of ≥ 30 on a numerical rating scale (0-100)

Exclusion Criteria:

* Starting a new daily prescription medication for the management of pain within 30 days prior to treatment session;
* Use of any injection therapy (e.g., tender or trigger point injections, steroid injections) for the management of pain within 2 weeks prior to the CATI;
* Starting occlusal appliance therapy within 30 days prior to CATI; d) history of facial trauma or orofacial surgery within 6 weeks prior to CATI;
* Active orthodontic treatment;
* Psychiatric hospitalization within one year prior to screening.
* Has known hypersensitivity to laser therapy.
* Currently being treated with chemotherapy or radiation therapy
* Has been treated with another investigational drug or treatment within 30 days prior to the Screening and Baseline Visit
* Is pregnant or nursing
* Anything that, in the opinion of the investigator, would place the participant at increased risk or preclude the participant's full compliance with or completion of the study

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 14 (Actual)
Dates: Start 2021-04-28 (Actual); Primary Completion 2022-12-16 (Actual); Study Completion 2022-12-16 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Margarete Ribeiro-Dasilva, DDS, MS, PhD, Principal Investigator — University of Florida
Locations (1):
- University of Florida, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One person was enrolled but withdrew prior to being assigned to a group which is why 14 people were enrolled but only 13 "started"
Period: Overall Study
Arm/Group | Active PBM | Sham PBM
Started | 7 | 6
Completed | 7 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Active PBM | Sham PBM | Total
Number analyzed (Participants) | 7 | 6 | 13
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 7 | 6 | 13
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 12
  Male | 1 | 0 | 1
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 7 | 5 | 12
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 7 | 6 | 13

OUTCOME MEASURES:

1. Primary Outcome: Pain Level Change With PBM Treatment Using a Numerical Rating Scale 0=no Pain and 100=the Most Intense Pain Imaginable
Description: Using a numerical rating scale (NRS) requires the patient to rate their pain on a defined scale 0=no pain and 100=the most intense pain imaginable to rate the average daily pain from Daily Pain & Symptom Dairy over one week prior to V1 will be compared to the average daily pain one week prior to V8.
Time Frame: Through study completion; an average of 10 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Active PBM | Sham PBM
Number analyzed (Participants) | 7 | 6
score on a scale | 5.8 (10.1) | 8.0 (18.0)

ADVERSE EVENTS:
Time Frame: each participant was assessed over their time in the study, about 3-6 weeks
Arm/Group | Active PBM | Sham PBM
All-Cause Mortality (participants affected / at risk) | 0/7 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/6
Other Adverse Events (participants affected / at risk) | 0/7 | 1/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Active PBM (N=7) | Sham PBM (N=6)
Discomfort around the face (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) — The participant experienced dry mouth, redness of the skin and general discomfort around the face.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-05-13): https://cdn.clinicaltrials.gov/large-docs/81/NCT04415281/Prot_SAP_002.pdf
  • Informed Consent Form (2022-06-21): https://cdn.clinicaltrials.gov/large-docs/81/NCT04415281/ICF_003.pdf